CLINICAL TRIAL: NCT00852553
Title: Neurohumoral Control of Intestinal Electrical and Mechanical Activity
Status: Completed | Type: Observational
Sponsor: University of California, Davis (Other)
Responsible Party: Sponsor
Other Study IDs: 200311379; 200311379-8
Record Dates: First submitted 2009-02-26; First posted 2009-02-27 (Estimated); Last update posted 2017-05-30 (Actual); Status verified 2017-05

CONDITIONS: Morbid Obesity
Keywords: intestinal; smooth; muscle; GI; motility
MeSH Terms: conditions — Obesity, Morbid

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — jejunum
Oversight: Data Monitoring Committee: No

SUMMARY:
A collaborative research project with Dr. Kathleen Keef (Department of Physiology, University of Nevada School of Medicine, Reno, Nevada) studying the role of putative neurotransmitters in human intestine.

DETAILED DESCRIPTION:
Segments of intestine from patients undergoing elective gastric bypass for morbid obesity or resections for non-obstructive neoplasms at the UC Davis Medical Center will be used. Samples will be taken from tissue normally removed and sent to Pathology or discarded. Full thickness segments of intestine (10 mm x 1 mm) will be prepared for recording either intracellular electrical activity or mechanical contraction. The effects of putative non-adrenergic, non-cholinergic neurotransmitters (e.g., nitric oxide) will be studied. The source of the tissue will not be identified either directly or indirectly through identifiers associated with the measured responses.

ELIGIBILITY:
Inclusion Criteria:

* All patients having elective bowel resection

Exclusion Criteria:

* Entire resected segment required for pathology
* Ischemic/necrotic disease

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All patients having elective bowel resections
Sampling Method: Non-Probability Sample
Enrollment: 45 (Actual)
Dates: Start 2003-02; Primary Completion 2012-02 (Actual); Study Completion 2012-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Neal W. Fleming, M.D., Ph.D., Principal Investigator — Professor
Locations (2):
- United States (2):
  - University of California, Davis Medical Center, Sacramento, California
  - University of Nevada School of Medicine, Reno, Nevada